CLINICAL TRIAL: NCT03835273
Title: Changes in Respiratory Function and Chest Wall Movement Following Oesophagectomy
Brief Title: Oesophagectomy and Chest Wall and Respiratory Function
Status: Recruiting | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 19SM5007
Record Dates: First submitted 2019-02-06; First posted 2019-02-08 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Esophageal Cancer; Esophagectomy; Respiratory Function Loss
Keywords: Esophagectomy; Motion capture; Respiratory; Oesophageal cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control group: Fourty control participants who have not received upper gastrointestinal surgery.
  Interventions: Other: 3D motion capture system; Other: Incentive spirometry; Other: Questionnaires
- Open surgery: Sixty patients who have undergone open removal of oesophagus more than one year ago.
  Interventions: Other: 3D motion capture system; Other: Incentive spirometry; Other: Questionnaires

INTERVENTIONS:
Other: 3D motion capture system — Small reflective markers and inertia measurement units will be placed on the chest of the patients using hypoallergenic adhesive and a motion capture system will pick up a 3D image via these markers non-invasively.
Other: Incentive spirometry — Incentive spirometry is a non-invasive device for assessment of pulmonary function.
Other: Questionnaires — Three validated, European Organisation for Research and Treatment of Cancer Quality-of-life Questionnaire Core 30 (EORTC QLQ-C30) and Oesophago-Gastric Module 25 (EORTC QLQ-OG25) and LASORS questionnaire.

SUMMARY:
Open surgery for esophageal cancer commonly involves large incisions in the chest, associated with a high rate of pulmonary complications (30-50%). Minimally invasive approach through keyhole surgery has been shown to reduce pulmonary infections by 20%. Enhanced recovery programmes are evidence-based protocols, developed to achieve early recovery after surgery with early mobilisation and chest physiotherapy and have been shown to reduce pulmonary complication rates as well. The investigators intend to objectively measure chest wall movement using 3D motion capture system as well as a wearable measurement system to monitor chest wall movement.

DETAILED DESCRIPTION:
The study population consists of 40 healthy volunteers who have not received upper gastrointestinal surgery and 60 patients treated with surgery more than one year ago (open approach). Chest wall movement will be measured using a 3D optical motion system and the investigators will establish if inertial measurement units placed strategically on the chest wall are able to quantify chest expansion and lung capacity. Data will be acquired during different breathing patterns and during use of an incentive spirometry. Pulmonary function tests will be undertaken in all patients and the investigators will also collect clinical data concerning health-related quality of life and other concomitant medical conditions. The target outcome of this study is to determine whether the 3D motion capture and wearable systems are reliable in the measurement of chest wall movement after surgical removal of esophagus and the validity and patient acceptability of wearable system, as well as the ability of distinguishing open and minimally invasive surgical approach. A tailored physiotherapy may be developed following this study in order to improve chest wall movement and objectively measure this using the wearable system. This can then be implemented in a clinical trial to provide the evidence base to for patient-tailored physiotherapy following major cancer surgery and to optimise the respiratory function.

ELIGIBILITY:
Inclusion Criteria:

* Exposure group:

  1. Patients treated more than a year ago with oesophagectomy for oesophageal cancer, by an open approach.
  2. Patients able to understand and retain the information provided, thereby being able to give informed consent for inclusion in this study.
* Control group:

  1. Healthy volunteers with no underlying respiratory disease and no history of upper gastrointestinal surgery.
  2. Individuals able to understand and retain the information provided, thereby being able to give informed consent for inclusion in this study.

Exclusion Criteria:

* Any participant who lacks capacity or is unable to provide informed consent.
* Any participant younger than 18 or older than 90 years of age.
* Any patient with evidence of cancer recurrence or on-going postoperative complication at more than one year following surgery for oesophageal cancer.
* Any pregnant participant.
* unable to or excluded from performing spirometry or respiratory muscle strength testing (non-invasive testing)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Three cohorts will be studied, equal in size. A total of 100 patients will be included in this study. One hundred patients who have undergone oesophagectomy for oesophageal cancer more than a year ago, 60 patients who have undergone open surgery and 40 healthy volunteers will be included as a control group with no underlying respiratory disease and no previous history of upper gastrointestinal surgery.
  Patients who have undergone oesophagectomy will be identified from existing databases by the direct care team of the patient. Healthy volunteers will be recruited from Imperial College through paper adverts.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-05-29 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Chest wall movement | Each participant will undergone one assessment during the study. The whole session, all procedures included, will last approximately 60 minutes.
  Evaluation of changes in chest wall movement in patients who have undergone oesophagectomy more than a year ago (open surgery) and in healthy control participants. Reflective markers will be placed on the chest wall of the participant and chest wall movement will be detected by a 3D motion capture system using these markers. In addition, inertia measurement units will be applied next to the markers. Chest wall movement will be assessed during normal breathing, take and hold a deep breath and whilst performing incentive spirometry.
Lung function | Each participant will undergone one assessment during the study. The whole session, all procedures included, will last approximately 60 minutes.
  Patients will be asked to perform incentive spirometry which is a non-invasive assessment of the lung function. Spirometry (tidal breathing, forced vital capacity) and respiratory muscle strength will be recorded for all participants.

SECONDARY OUTCOMES:
Health-related Quality of Life in cancer patients | Each participant will undergone one assessment during the study. The whole session, all procedures included, will last approximately 60 minutes.
  All participants will be asked to fill in a validated questionnaire, the European Organisation for Research and Treatment of Cancer Quality-of-life Questionnaire Core 30 (EORTC QLQ-C30) for assessment of their current quality of life. The QLQ-C30 includes 5 functional scales, 3 symptom scales, a global health status/QoL scale, and 6 single items. Items 1 to 28 have a four-point scale response, namely 'Not at all' (point 1), 'A little', 'Quite a bit' and 'Very much' (point 4). The last 2 items have a seven-point scale for assessment of the overall health and overall quality of life, being 'Very poor' (point 1) to 'Excellent (points 7). Higher scores in the function and global quality of life scales represent better levels outcome, whilst higher scores in symptom scales represent presence of more symptoms. Similarly, the EORTC QLQ-25 comprises of questionnaires to assess the quality of life. LASORS questionnaire assesses the long-term deficits in quality of life in this population.
Health-related Quality of Life in patients with tumours of the oesophagus, oesophago-gastric junction or stomach | Each participant will undergone one assessment during the study. The whole session, all procedures included, will last approximately 60 minutes.
  All participants will be asked to fill in a validated questionnaire, European Organisation for Research and Treatment of Cancer Quality-of-life Questionnaire Oesophago-Gastric Module 25 (EORTC QLQ-OG25) for assessment of their current quality of life. The QLQ-OG25 has six symptom scales (dysphagia, eating restrictions, reflux, odynophagia, pain and discomfort, and a scale assessing anxiety) and 10 single items relevant to patients undergoing palliative or potentially curative treatments and follow-up for upper gastrointestinal cancer. All items have four-point scale, namely 'Not at all' (point 1), 'A little', 'Quite a bit' and 'Very much' (point 4). Higher scores in symptom scales represent presence of more symptoms.

OTHER OUTCOMES:
Usability and acceptability of the measuring device | Each participant will undergone one assessment during the study. The whole session, all procedures included, will last approximately 60 minutes.
  All participants will be asked to fill in a satisfaction questionnaire regarding the usability and acceptability of the 3D motion capture system. This questionnaire includes a total of 10 items assessing the usability and acceptability of the 3D motion capture system. Each item has a five-point Likert scale response, with 'Strongly disagree' (point 1), 'Disagree', 'Neutral', 'Agree' and 'Strongly agree' (point 5). Higher scores correspond with better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Sheraz R Markar, Dr, Principal Investigator — Imperial College London
Locations (1):
- Charing Cross Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shirinzadeh A, Talebi Y. Pulmonary Complications due to Esophagectomy. J Cardiovasc Thorac Res. 2011;3(3):93-6. doi: 10.5681/jcvtr.2011.020. Epub 2011 Aug 20. PMID 24250962
- [Background] Nagawa H, Kobori O, Muto T. Prediction of pulmonary complications after transthoracic oesophagectomy. Br J Surg. 1994 Jun;81(6):860-2. doi: 10.1002/bjs.1800810622. PMID 8044603
- [Background] Biere SS, van Berge Henegouwen MI, Maas KW, Bonavina L, Rosman C, Garcia JR, Gisbertz SS, Klinkenbijl JH, Hollmann MW, de Lange ES, Bonjer HJ, van der Peet DL, Cuesta MA. Minimally invasive versus open oesophagectomy for patients with oesophageal cancer: a multicentre, open-label, randomised controlled trial. Lancet. 2012 May 19;379(9829):1887-92. doi: 10.1016/S0140-6736(12)60516-9. Epub 2012 May 1. PMID 22552194
- [Background] Kubo N, Ohira M, Yamashita Y, Sakurai K, Toyokawa T, Tanaka H, Muguruma K, Shibutani M, Yamazoe S, Kimura K, Nagahara H, Amano R, Ohtani H, Yashiro M, Maeda K, Hirakawa K. The impact of combined thoracoscopic and laparoscopic surgery on pulmonary complications after radical esophagectomy in patients with resectable esophageal cancer. Anticancer Res. 2014 May;34(5):2399-404. PMID 24778050
- [Background] Schmidt HM, El Lakis MA, Markar SR, Hubka M, Low DE. Accelerated Recovery Within Standardized Recovery Pathways After Esophagectomy: A Prospective Cohort Study Assessing the Effects of Early Discharge on Outcomes, Readmissions, Patient Satisfaction, and Costs. Ann Thorac Surg. 2016 Sep;102(3):931-939. doi: 10.1016/j.athoracsur.2016.04.005. Epub 2016 Jun 7. PMID 27283109
- [Background] Li C, Ferri LE, Mulder DS, Ncuti A, Neville A, Lee L, Kaneva P, Watson D, Vassiliou M, Carli F, Feldman LS. An enhanced recovery pathway decreases duration of stay after esophagectomy. Surgery. 2012 Oct;152(4):606-14; discussion 614-6. doi: 10.1016/j.surg.2012.07.021. Epub 2012 Sep 1. PMID 22943844
- [Background] Aaronson NK, Ahmedzai S, Bergman B, Bullinger M, Cull A, Duez NJ, Filiberti A, Flechtner H, Fleishman SB, de Haes JC, et al. The European Organization for Research and Treatment of Cancer QLQ-C30: a quality-of-life instrument for use in international clinical trials in oncology. J Natl Cancer Inst. 1993 Mar 3;85(5):365-76. doi: 10.1093/jnci/85.5.365. PMID 8433390
- [Background] Lagergren P, Fayers P, Conroy T, Stein HJ, Sezer O, Hardwick R, Hammerlid E, Bottomley A, Van Cutsem E, Blazeby JM; European Organisation for Research Treatment of Cancer Gastrointestinal and Quality of Life Groups. Clinical and psychometric validation of a questionnaire module, the EORTC QLQ-OG25, to assess health-related quality of life in patients with cancer of the oesophagus, the oesophago-gastric junction and the stomach. Eur J Cancer. 2007 Sep;43(14):2066-73. doi: 10.1016/j.ejca.2007.07.005. Epub 2007 Aug 15. PMID 17702567